CLINICAL TRIAL: NCT04737668
Title: Virtual Reality During Intrathecal Pump Refills in Children: a Randomised Controlled Trial With Crossover Design
Brief Title: Virtual Reality During Intrathecal Pump Refills in Children
Acronym: VAMPIRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Moens Maarten (Other)
Responsible Party: Sponsor-Investigator, Moens Maarten, principal investigator, Universitair Ziekenhuis Brussel
Organization: Universitair Ziekenhuis Brussel (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: VAMPIRE
Record Dates: First submitted 2021-01-26; First posted 2021-02-04 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Cerebral Palsy
Keywords: Virtual Reality
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual care (Other): Pump refill will be performed as usual.
  Interventions: Other: Intrathecal pump refill
- Virtual Reality (Other): Children will play a commercially available VR game during pump refill
  Interventions: Other: Intrathecal pump refill with Virtual Reality
- Distraction (Other): Children will watch a commercial 360° music video on YouTube during pump refill
  Interventions: Other: Intrathecal pump refill with distraction

INTERVENTIONS:
Other: Intrathecal pump refill with Virtual Reality — VR game
  Arms: Virtual Reality
Other: Intrathecal pump refill with distraction — Video
  Arms: Distraction
Other: Intrathecal pump refill — daily routine care for pump refill
  Arms: Usual care

SUMMARY:
The aim of the current study is to explore the effect of virtual reality on pain in children who undergo an intrathecal pump refill compared to usual care and distraction.

DETAILED DESCRIPTION:
Virtual reality (VR) is a technological rehabilitation tool that allows the user to experience the interaction with a computer-generated environment. It may provide some advantages over conventional care: it allows the simulation of realistic environments and patients feel more motivated by this kind of virtual environment. VR constitutes an enriched environment with augmented multiple sensory feedbacks (auditory, visual, tactile VR enriched environment) that has already shown some efficiency in reducing chronic pain. There is mounting evidence from acute pain conditions, such as wound care, that VR could play a role as an additional treatment method to relieve pain A possible explanation for its mechanism of action is provided by "the gate-theory of attention". VR reduces the perception of pain by diverting attention away from the pain. Most children experience pain and fear when receiving a medical treatment; two feelings which are closely related and affecting one another. Moreover, children often describe procedures involving needles as the most stressful portion of the hospital experience. Children who have been implanted with an intrathecal baclofen (ITB) pump, need to come to the hospital for a refill approximately every 3 months, depending on the exact dose. During the refill, the physician places a needle directly into the reservoir to refill the pump. To alleviate the pain and fear with these refill procedures, it is hypothesized that VR could alleviate pain and make these refills more feasible. Therefore, the aim of this study is to evaluate whether VR is reducing pain during a refill procedure, in children receiving intrathecal drug delivery compared to usual care.

ELIGIBILITY:
Inclusion Criteria:

* Children with cerebral palsy between 8 and 16 years who have an implanted pump for intrathecal drug delivery
* Child and parents have been informed of the study procedures and have given written informed consent
* Child and parents willing to comply with study protocol
* Child and parents are able to speak Dutch/French (questionnaires)
* Cognitive and language functioning enabling communication between the physician/researcher and the child

Exclusion Criteria:

* Children with susceptibility to motion sickness or cyber-sickness
* Children with susceptibility to claustrophobia
* History of seizures/epilepsia

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2021-02-10 (Actual); Primary Completion 2022-01-26 (Actual); Study Completion 2022-01-26 (Actual)

PRIMARY OUTCOMES:
Pain intensity | Through study completion, an average of 6 months.
  Pain intensity will be assessed with the Wong-Baker FACES scale in children, parents, physician and researcher, to evaluate differences in the 3 conditions (usual refill, refill with VR and refill with distraction).

SECONDARY OUTCOMES:
Procedural pain | Through study completion, an average of 6 months.
  Procedural pain during refill is assessed with the Face, Legs, Activity, Cry, Consolability scale.
Fear | Through study completion, an average of 6 months.
  The degree of fear will be measured using the Child Fear Scale, based on reporting from the child and parent.
Anxiety | Through study completion, an average of 6 months.
  The Children's Anxiety Meter (CAM) will be used to measure anxiety. This scale will be filled in by children and parents.
Statisfaction | Through study completion, an average of 6 months.
  The statisfaction will be evaluated by two questions, scoring on a 5-point Likert agreement scale, by the children, parents and physician after the refill with VR and after the refill with distraction.
Adverse events | Through study completion, an average of 6 months.
  The incidence of adverse events (nausea, vomiting, motion sickness, dizziness, seizure) will be evaluated after the refill with VR.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitair Ziekenhuis Brussel, Jette, Belgium